CLINICAL TRIAL: NCT06676072
Title: Safety and Effectiveness of the TactiFlex SE Catheter and Volt Pulsed Field Ablation (PFA) Generator in Subjects With Paroxysmal Atrial Fibrillation
Brief Title: A Study of the TactiFlex SE Catheter and Volt PFA Generator in Subjects With PAF:
Acronym: FlexPulse IDE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-CIP-10520
Record Dates: First submitted 2024-11-04; First posted 2024-11-06 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation (AF); Atrial Arrhythmia; Paroxysmal AF; Drug Refractory Paroxysmal Atrial Fibrillation
Keywords: Symptomatic, recurrent, drug refractory PAF; Atrial Fibrillation; Paroxysmal AF; Pulsed Field Ablation; Radio Frequency; PFA
MeSH Terms: conditions — Atrial Fibrillation; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TactiFlex Ablation catheter (Experimental): A single use catheter that is designed to facilitate electrophysiological mapping of the heart chambers and to transmit RF current or PFA therapy to the catheter's flexible tip electrode for intracardiac ablation purposes.
  Interventions: Device: PFA Ablation catheter

INTERVENTIONS:
Device: PFA Ablation catheter — Deliver RF and/or PF energy using the TactFlex PFA system

SUMMARY:
The objective of this clinical study is to demonstrate that ablation with the TactiFlex SE Ablation catheter, in conjunction with a compatible pulsed field ablation (PFA) and/or radio frequency (RF) generator, is safe and effective for the treatment of symptomatic, recurrent, drug refractory paroxysmal atrial fibrillation (PAF).

DETAILED DESCRIPTION:
This is a pre-market, prospective, single-arm, non-randomized, multicenter clinical study to demonstrate safety and effectiveness for the treatment of symptomatic, recurrent, drug-refractory PAF.

ELIGIBILITY:
Inclusion Criteria:

1. Documented symptomatic paroxysmal atrial fibrillation (PAF). Documentation requirements are as follows:

   1. Physician's note indicating recurrent self-terminating AF with ≥ 2 episodes of PAF within the 6 months prior to enrollment AND
   2. One electrocardiographically documented PAF episode within 12 months prior to enrollment.

   NOTE: Documented evidence of the AF episode must either be continuous AF on a 12-lead ECG or include at least 30 seconds of continuous AF from another ECG device.
2. Plans to undergo a catheter ablation procedure due to symptomatic PAF and is refractory, intolerant, or contraindicated to at least one Class I-IV AAD medication
3. At least 18 years of age
4. Able and willing to comply with all trial requirements including pre- procedure, post-procedure, and follow-up testing and requirements
5. Informed of the nature of the trial, agreed to its provisions, and has provided written informed consent as approved by the Institutional Review Board/Ethics Committee (IRB/EC) of the respective clinical trial site.

Exclusion Criteria:

1. Previously diagnosed persistent or long-standing persistent atrial fibrillation (Continuous AF greater than 1 year in duration)
2. Arrhythmia due to reversible causes including thyroid disorders, acute alcohol intoxication, electrolyte imbalance, severe untreated sleep apnea, and other major surgical procedures in the preceding 90 days
3. Known presence of cardiac thrombus
4. Left atrial diameter (LAD) > or equal to 5.0 cm (anteroposterior diameter) within 180 days prior to the index procedure
5. Left ventricular ejection fraction (LVEF) < or equal to 35% as assessed with echocardiography or computerized tomography (CT) within 180 days prior to the index procedure
6. New York Heart Association (NYHA) class III or IV heart failure
7. Body mass index > or equal to 40 kg/m2
8. Pregnant or nursing
9. Patients who have had a ventriculotomy or atriotomy within the preceding 28 days of procedure
10. Myocardial infarction (MI), acute coronary syndrome, percutaneous coronary intervention (PCI), or valve or coronary bypass grafting surgery within preceding 90 days
11. Stroke or TIA (transient ischemic attack) within the last 90 days
12. Heart disease in which corrective surgery is anticipated within 180 days after procedure
13. History of blood clotting or bleeding abnormalities including thrombocytosis, thrombocytopenia, bleeding diathesis, or suspected anti- coagulant state
14. Contraindication to long-term anti-thromboembolic therapy
15. Patient unable to receive heparin or an acceptable alternative to achieve adequate anticoagulation
16. Known sensitivity to contrast media (if needed during the procedure) that cannot be controlled with pre-medication
17. Previous left atrial surgical or left atrial catheter ablation procedure (including left atrial appendage (LAA) closure device)
18. Plans to have an LAA closure device implanted during the follow-up period
19. Presence of any condition that precludes appropriate vascular access
20. Severe mitral regurgitation (regurgitant volume ≥ 60 mL/beat, regurgitant fraction ≥ 50%, and/or effective regurgitant orifice area ≥ 0.40cm2)
21. Previous tricuspid or mitral valve replacement or repair
22. Patients with prosthetic valves
23. Patients with a myxoma
24. Patients with an interatrial baffle or patch as the transseptal puncture could persist and produce an iatrogenic atrial shunt
25. Stent, constriction, or stenosis in a pulmonary vein
26. Rheumatic heart disease
27. Hypertrophic cardiomyopathy
28. Active systemic infection
29. Renal failure requiring dialysis
30. Severe pulmonary disease (e.g., restrictive pulmonary disease, constrictive or chronic obstructive pulmonary disease) or any other disease or malfunction of the lungs or respiratory system that produces severe chronic symptoms
31. Presence of an implantable therapeutic cardiac device including permanent pacemaker, biventricular pacemaker, or any type of implantable cardiac defibrillator (with or without biventricular pacing function) or planned implant of such a device for any time during the follow-up period. Presence of an implantable loop recorder is acceptable as long as it is removed prior to insertion of the investigational device.
32. Patient is currently participating in another clinical trial or has participated in a clinical trial within 30 days prior to screening that may interfere with this clinical trial without pre-approval from this study Sponsor
33. Unlikely to survive the protocol follow up period of 12 months
34. Presence of other medical, anatomic, comorbid, social, or psychological conditions that, in the investigator's opinion, could limit the subject's ability to participate in the clinical investigation or to comply with follow-up requirements, or impact the scientific soundness of the clinical investigation results.
35. Individuals without legal authority
36. Individuals unable to read or write

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Estimated)
Dates: Start 2024-11-22 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects experiencing a device and/or procedure-related serious adverse event with onset within 7 days of any ablation procedure (index or repeat procedure performed 0-90 days post initial procedure). | 7 days
Freedom from documented (symptomatic or asymptomatic) AF/AFL/AT episodes of greater than 30 seconds duration that are documented by protocol-specified 12-lead ECG, TTM or Holter monitor (HM) devices after the index ablation procedure | 12 months

SECONDARY OUTCOMES:
Symptomatic Effectiveness | 12 months
  Freedom from documented symptomatic AF/AF/AT episodes of greater than 30 seconds duration that are documented by protocol-specific 12-lead ECG, TTM or Holter monitor devices after the index ablation procedure.
AAD-Free Effectiveness | 12 months
  Freedom from documented (symptomatic or asymptomatic) AF/AFL/AT episodes of > 30 seconds duration that are documented by protocol-specific 12-lead ECG, TTM, or Holter monitor after the index ablation procedure. Any use of Class I or III antiarrythmic drugs after the 90-day blanking period will count as a therapy failure in the analysis

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kammer, Study Director — Abbott Medical Devices
Locations (32):
- United States (29):
  - HonorHealth, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Stanford University Medical Center, Stanford, California
  - South Denver Cardiology Associates PC, Littleton, Colorado
  - HCA Florida Mercy Hospital, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - Tallahassee Research Institute, Tallahassee, Florida
  - Piedmont Athens Regional Medical Center, Athens, Georgia
  - Loyola University Medical Center, Maywood, Illinois
  - Kansas City Cardiac Arrhythmia Research Foundation, Overland Park, Kansas
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Henry Ford Providence Southfield Hospital, Southfield, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - The Heart Rhythm Center of MS, Gulfport, Mississippi
  - Bryan Heart Medical Center, Lincoln, Nebraska
  - NYU Langone Health, New York, New York
  - New York Presbyterian Hospital/Cornell University, New York, New York
  - Duke University Medical Center, Durham, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Tristar Centennial Medical Center, Nashville, Tennessee
  - Vanderbilt Heart & Vascular Institute, Nashville, Tennessee
  - Texas Cardiac Arrhythmia, Austin, Texas
  - Ocelot Medical Research Group, Dallas, Texas
  - Medical City Fort Worth, Fort Worth, Texas
  - Houston Methodist The Woodlands Hospital, Shenandoah, Texas
  - Virginia Commonwealth University, Richmond, Virginia
  - The Heart Institute at Virginia Mason, Seattle, Washington
- KH Wiener Neustadt, Wiener Neustadt, L Austr, Austria
- Vilnius University Hospital Santariskiu Klinikos, Vilnius, Dzukija, Lithuania
- Erasmus Medical Center - Thoraxcenter, Rotterdam, S Holln, Netherlands

IPD SHARING:
Plan to Share IPD: No